CLINICAL TRIAL: NCT03018509
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of JTE-451 Administered for 4 Weeks in Subjects With Active Plaque Psoriasis
Brief Title: Study to Evaluate Safety,Tolerability,Pharmacodynamics & Pharmacokinetics of JTE-451 in Active Plaque Psoriasis Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AE451-X-16-003
Record Dates: First submitted 2017-01-06; First posted 2017-01-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Plaque Psoriasis; Psoriasis; Skin Diseases
Keywords: JTE-451; psoriasis
MeSH Terms: conditions — Psoriasis; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- JTE-451 Dose 1 (Experimental): JTE-451 dose 1 for 28 days
  Interventions: Drug: JTE-451
- JTE-451 Dose 2 (Experimental): JTE-451 dose 2 for 28 days
  Interventions: Drug: JTE-451
- JTE-451 Dose 3 (Experimental): JTE-451 dose 3 for 28 days
  Interventions: Drug: JTE-451
- JTE-451 Dose 4 (Experimental): JTE-451 dose 4 for 28 days
  Interventions: Drug: JTE-451
- Placebo (Experimental): Placebo for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JTE-451 — Active drug tablets containing JTE-451
  Arms: JTE-451 Dose 1; JTE-451 Dose 2; JTE-451 Dose 3; JTE-451 Dose 4
Drug: Placebo — Placebo tablets identical in appearance to the active drug tablets
  Arms: Placebo

SUMMARY:
Study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamic effect of JTE-451 administered for 4 weeks in subjects with active plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of two psoriatic plaques (i.e., one clinical target lesion and one biopsy target lesion).
* Each of the two target lesions must have a psoriatic lesion severity sum (PLSS) of ≥6
* Body mass index (BMI) of 18 to 38 kg/m2 (inclusive)

Exclusion Criteria:

* Prior exposure to >2 systemic biologic agents and/or small molecules including investigational therapies for the treatment of psoriasis or have not discontinued systemic biologic agents and/or small molecules anti-psoriasis therapy including investigational therapies due to lack of efficacy;
* Subjects with significant health problems, other than having plaque psoriasis (as determined by medical history, physical examination, chest X-ray, vital signs and 12-lead ECG) that could either interfere with study evaluations or place subject at undue risk;
* Presence of erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis at Visit 1;
* Conditions (e.g., clinically-significant eczema or severe acne in the target lesion area) that would interfere with study evaluations;
* Positive quantiFERON®-TB Gold test, negative chest X-ray findings for tubercle bacillus (TB) or lack any other evidence of active or latent TB;
* History of a clinically-significant infection (e.g., required oral antimicrobial therapy) within 4 weeks prior to Visit 2;
* Subjects who do not have clinical laboratory test results within the normal reference ranges (i.e., are deemed not to be clinically significant) or clinically not acceptable to the Investigator;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-12; Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 4 weeks
Percent change from baseline in the clinical target PLSS | Weeks 1, 2, 3 and 4
Percent change from baseline in the clinical target lesion erythema | Weeks 1, 2, 3 and 4
Percent change from baseline in the clinical target lesion induration | Weeks 1, 2, 3 and 4
Percent change from baseline in the clinical target lesion scaling | Weeks 1, 2, 3 and 4
Change from baseline in the clinical target lesion sPGA score | Weeks 1, 2, 3 and 4
Number of subjects with clinical target lesion sPGA scores of 0 or 1 | Week 1
Number of subjects with clinical target lesion sPGA scores of 0 or 1 | Week 2
Number of subjects with clinical target lesion sPGA scores of 0 or 1 | Week 3
Number of subjects with clinical target lesion sPGA scores of 0 or 1 | Week 4
Number of subjects with at least a 2-point improvement in sPGA score | Baseline to Week 4
Trough concentration during multiple dosing prior to next dose (Ctrough) | Weeks 1, 2, 3 and 4

CONTACTS AND LOCATIONS:
Locations (5):
- Canada (5):
  - Surrey, British Columbia
  - Markham, Ontario
  - Peterborough, Ontario
  - Richmond Hill, Ontario
  - Waterloo, Ontario

IPD SHARING:
Plan to Share IPD: No